CLINICAL TRIAL: NCT00260078
Title: Intensive Pharmacokinetic Studies of Antiretroviral Drug Combinations in Children
Brief Title: Blood Levels of Anti-HIV Drugs Used in Combination Regimens in HIV Infected Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1058; PACTG 1058; IMPAACT P1058; 10050 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2016-07

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Pharmacokinetics; PK
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Darunavir; efavirenz; Nevirapine; Ritonavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- D (Experimental): TDF and EFV or NVP throughout study
  Interventions: Drug: Efavirenz; Drug: Nevirapine; Drug: Tenofovir disoproxil fumarate; Procedure: Pharmacokinetic Study
- E (Experimental): TDF and DRV with or without EFV throughout study
  Interventions: Drug: Darunavir; Drug: Efavirenz; Drug: Ritonavir; Drug: Tenofovir disoproxil fumarate; Procedure: Pharmacokinetic Study
- F (Experimental): TDF and ATV and RTV with or without EFV throughout study
  Interventions: Drug: Atazanavir; Drug: Efavirenz; Drug: Ritonavir; Drug: Tenofovir disoproxil fumarate; Procedure: Pharmacokinetic Study

INTERVENTIONS:
Drug: Atazanavir — 200 mg to 400 mg orally daily
  Other Names: ATV
  Arms: F
Drug: Darunavir — 300 mg or 600 mg orally twice daily
  Other Names: DRV
  Arms: E
Drug: Efavirenz — Dosage dependent on participant
  Other Names: EFV
Drug: Nevirapine — Dosage dependent on participant
  Other Names: NVP
  Arms: D
Drug: Ritonavir — 50 mg or 100 mg orally twice daily
  Other Names: RTV
  Arms: E; F
Drug: Tenofovir disoproxil fumarate — 300 mg orally daily
  Other Names: TDF
Procedure: Pharmacokinetic Study — Intensive PK study will occur at least once. This will require a 24-hour inpatient visit.
  Other Names: PK Study

SUMMARY:
Limited data exist about combination anti-HIV treatment regimens in children, including how those drugs are cleared by the body in children. The purpose of this study is to measure the blood levels of the following combinations of anti-HIV drugs in HIV infected chilren: tenofovir disoproxil fumurate (TDF) and efavirenz (EFV) or nevirapine (NVP); TDF and darunavir (DRV) with or without EFV; and TDF and ritonavir (RTV) with or without EFV.

DETAILED DESCRIPTION:
Because all of the available non-nucleoside reverse transcriptase inhibitors (NNRTIs) and protease inhibitors (PIs) are metabolized by and affect hepatic cytochrome enzymes, combinations of two or more of these drugs produce complex pharmacokinetic (PK) interactions. However, little data exist regarding PK of anti-HIV drug combinations in the pediatric population. The purpose of this study is to assess steady-state PK of the following anti-HIV regimens: TDF and EFV or NVP; TDF and DRV with or without EFV; and TDF and RTV with or without EFV. In addition, this study will evaluate how age, length of treatment, adverse effects, and genes affect children's response to different anti-HIV combinations.

This study will last between 1 and 7 weeks. Participants in this study will be grouped based on the treatment regimen they are receiving or about to initiate. There are three groups in this study. Group D participants will receive TDF and EFV or NVP; Group E participants will receive TDF and DRV with or without EFV; and Group F participants will receive TDF and RTV with or without EFV. The inclusion of EFV or NVP will be dependent on each participant's prescribed regimen. Participants within each group will be stratified by age and how long they have been receiving their anti-HIV regimens. Antiretrovirals will not be provided by this study.

Most participants will have two study visits. The first visit will occur at study entry. Medical history, a physical exam, and blood collection will occur. The second visit will occur within 35 days of study entry and will take approximately 24 hours. Blood collection for PK studies, a physical exam, and medical history will be done at this visit. Urine collection will occur at all visits for female participants.

Participants will undergo PK testing at least 14 days after initiating their study regimens. Participants will be given a dose of their anti-HIV medications with food. A blood sample will be taken before dosing. Blood samples will also be taken at 1, 2, 4, 6, 8, 12, and 24 hours after dosing. Participants in Groups E and F may need to repeat PK testing within 6 weeks of initial PK testing at the discretion of the investigator.

ELIGIBILITY:
Note: The original Groups A, B, and C have been removed, and Groups D, E, and F have been added per protocol amendment dated 11/16/07.

Inclusion Criteria:

* HIV infected
* Currently receiving or about to initiate one of the following anti-HIV regimens: TDF with EFV or NVP, TDF and DRV/r with or without EFV, or TDF with ATV/r with or without EFV
* Body surface area at least 0.85 m2
* Parent or guardian willing and able to provide signed informed consent
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Liver disease that may affect the metabolism of study drugs
* Certain abnormal laboratory values
* Require certain medications
* Treatment with any anti-HIV or nonantiretroviral drug that could interact with drugs under PK study in the 14 days prior to study entry
* Any clinical or laboratory toxicity of Grade 4 or higher at screening. More information on this criterion can be found in the protocol.
* Pregnant or breastfeeding

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Predosage concentration (C0 and C12) and area under the concentration-time curve (AUC) | Over the dosing interval

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer King, PharmD, Study Chair — Department of Pharmacology and Toxicology, University of Alabama at Birmingham; Ram Yogev, MD, Study Chair — Section of Pediatrics and Maternal HIV Infection, Children's Memorial Hospital, Northwestern University Medical School
Locations (23):
- United States (21):
  - Usc La Nichd Crs, Alhambra, California
  - University of California, UC San Diego CRS, La Jolla, California
  - Miller Children's Hosp. Long Beach CA NICHD CRS, Long Beach, California
  - Harbor UCLA Medical Ctr. NICHD CRS, Torrance, California
  - Connecticut Children's Med. Ctr., Hartford, Connecticut
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Ann & Robert H. Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - Univ. of Maryland Baltimore NICHD CRS, Baltimore, Maryland
  - Johns Hopkins Univ. Baltimore NICHD CRS, Baltimore, Maryland
  - Children's Hosp. of Boston NICHD CRS, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - Rutgers - New Jersey Medical School CRS, Newark, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - Nyu Ny Nichd Crs, New York, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS, The Bronx, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
  - Seattle Children's Hospital CRS, Seattle, Washington
- Puerto Rico (2):
  - University of Puerto Rico Pediatric HIV/AIDS Research Program CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Kiser JJ, Fletcher CV, Flynn PM, Cunningham CK, Wilson CM, Kapogiannis BG, Major-Wilson H, Viani RM, Liu NX, Muenz LR, Harris DR, Havens PL; Adolescent Trials Network for HIV/AIDS Interventions. Pharmacokinetics of antiretroviral regimens containing tenofovir disoproxil fumarate and atazanavir-ritonavir in adolescents and young adults with human immunodeficiency virus infection. Antimicrob Agents Chemother. 2008 Feb;52(2):631-7. doi: 10.1128/AAC.00761-07. Epub 2007 Nov 19. PMID 18025112
- [Background] Hazra R, Gafni RI, Maldarelli F, Balis FM, Tullio AN, DeCarlo E, Worrell CJ, Steinberg SM, Flaherty J, Yale K, Kearney BP, Zeichner SL. Tenofovir disoproxil fumarate and an optimized background regimen of antiretroviral agents as salvage therapy for pediatric HIV infection. Pediatrics. 2005 Dec;116(6):e846-54. doi: 10.1542/peds.2005-0975. Epub 2005 Nov 15. PMID 16291735